CLINICAL TRIAL: NCT06292806
Title: Assessment of Ovarian Responsiveness Through AMH/AFC and Inhibin B/AFC Ratio
Brief Title: Inhibin B/AFC Ratio for Ovarian Response
Status: Not yet recruiting | Type: Observational
Sponsor: Insemine Humen Reproduction Centre (Network)
Responsible Party: Sponsor
Other Study IDs: 001-2024
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: IVF; Infertility, Female; Ovulation Disorder
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: FSH-R — controlled ovarian stimulation for IVF

SUMMARY:
Ovarian response to gonadotropin stimulation plays a major role in the success of in vitro fertilization (IVF). Anti-müllerian hormone (AMH), inhibin B, and antral follicle count (AFC) are ovarian reserve markers and also predictors of the ovarian response, as they correlate with the number of oocytes retrieved. Ovarian responsiveness can also be assessed through the Follicular Output Rate (FORT), which evaluates the proportion of follicles that developed during stimulation by the ratio of PFC (preovulatory follicle count) to AFC. FORT highlights that some follicles do not respond to the FSH; therefore, this project proposes an endocrinological approach to this issue by relating AFC to inhibin B and AMH ㅡ hormones produced by granulosa cells, but at different stages of folliculogenesis and with endocrine and paracrine functions, respectively. The inhibin B/AFC and AMH/AFC ratios correlated with FORT and the number of oocytes retrieved may help elucidate the mechanisms involved in follicular responsiveness.

A prospective cohort study will be conducted with patients of the Insemine Center for Human Reproduction. Antral follicle count and AMH measurement will be performed before IVF cycle initiation, and inhibin B measurement will be carried out on a blood sample collected on the fifth day of ovarian stimulation. The primary outcomes will be the Follicular Output Rate (FORT) and the number of oocytes retrieved. Secondary outcomes include the number of metaphase II oocytes, oocyte quality, fertilization rate and embryo quality.

ELIGIBILITY:
Inclusion Criteria:

* first IVF;
* without severe male factor involved.

Exclusion Criteria:

* Patients with endometrioma;
* ovarian cyst;
* AMH < 0.5 ng/ml;
* increased serum TSH (thyroid-stimulating hormone) or prolactin levels;
* endocrinopathies;
* previous oophorectomy;
* failure to visualize one of the ovaries on ultrasound.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Follicle counting (AFC) will be performed prior to the administration of gonadotropins. For ovarian stimulation, a flexible protocol will be used with a GnRH antagonist (gonadotropin-releasing hormone) and doses of 150-300 IU of recombinant FSH administered daily. Follicular growth will be monitored by ultrasound and hCG (human chorionic gonadotropin) will be administered when two or more follicles reach 17 mm in diameter; In this last ultrasound, the pre-ovulatory follicle count (PFC) will be performed to calculate the FORT. Ovarian puncture will be performed 36 hours after hCG administration. On the fifth day of induction, a blood sample will be collected from the patient for subsequent inhibin B measurement by enzyme-linked immunosorbent assay (ELISA). These samples will be stored at the Insemine Human Reproduction Center
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
serum Inhibin B levels | Day 1 and Day 5 of controlled ovarian stimulation
serum Anti Mullerian Hormone levels | Day 1 and Day 5 of controlled ovarian stimulation

IPD SHARING:
Plan to Share IPD: Undecided